CLINICAL TRIAL: NCT04291755
Title: Development and Analysis of a Sample Bank (Blood, Urine, and Stool) for Cancer Patients, Enabling the Systematic Study of the Effect of Blood, Urinary Tract, and Gut Microbiomes on Response to Treatment
Brief Title: Development and Analysis of a Stool Bank for Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Persephone Biosciences (Industry)
Collaborators: Pharm-Olam International (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-002
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Colorectal
Keywords: Non-small cell lung cancer; immunotherapy; checkpoint inhibitor; pembrolizumab; nivolumab; ipilimumab; microbiome
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — pembrolizumab; Nivolumab; Ipilimumab; tocilizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, blood, and urine specimens from each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Checkpoint inhibitor therapy: Patients will be administered a checkpoint inhibitor therapy, including but not limited to pembrolizumab, nivolumab, ipilimumab, and atlizumab, at the standard dosing regimen prescribed by their physician. Stool, blood, and urine samples will be collected from patients prior to start of treatment, and at 4 more timepoints over the next 12 months.
  Interventions: Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Pembrolizumab Injection — Any checkpoint inhibitor is acceptable
  Other Names: nivolumab, ipilimumab, atlizumab

SUMMARY:
This study is aimed at understanding the impact of gut microbiota on efficacy of cancer therapies, in particular checkpoint inhibitors, and using the resulting information to design microbial immunotherapies. Although animal models are of use to determine the influences of gut and other microbiota on cancer treatment modalities, they are limited due to differences between mouse and human physiology and immunology, as well as the inherent differences in gut microbial populations between the two mammalian organisms. Therefore, samples obtained as donations from human subjects undergoing cancer treatment are of great value for the identification and determination of bacteria and their metabolic processes that are involved in the successful cure and remission of cancer by checkpoint inhibitor therapies.

The objective of this study is to collect 3 samples each of blood, urine, and stool in subjects with cancer. This is a non-interventional, 2 site study in 100 people who are undergoing any type of cancer immunotherapy. Subjects who meet the entry criteria will provide 5 samples each of blood, urine, and stool over a 12-month period.

DETAILED DESCRIPTION:
A growing body of evidence indicates that the composition of the gut microbiome can influence the efficacy of cancer drugs. For example, it has recently been demonstrated that the presence of certain microbes in the gut is correlated with better responsiveness to the new immunotherapy drugs known as checkpoint inhibitors. Providing these particular microbes as a co-therapy may be a way to improve the overall success rate of these drugs. However, very little is currently known about the mechanisms involved in these observed positive effects.

In order to systematically identify how the presence or absence of particular microbes modulates responsiveness to checkpoint inhibitors and other immunotherapy drugs, Persephone Biome is building a biobank comprised of donated samples from a diversity of cancer patients undergoing various anti-cancer treatments. These samples will be analyzed using metabolic models and machine learning approaches to identify microbial species, gene functions, and metabolic pathways that are associated with efficacy and toxicity of treatments. Ultimately, these data will facilitate the development of live biotherapeutics as co-therapies to various cancer drugs.

This is a non-interventional, 2 site study in 100 subjects who are undergoing any type of cancer immunotherapy. It is preferred that enrollment is balanced by sex; however, it is not required. Subjects who meet the entry criteria will provide 5 samples each of blood, urine, and stool over a 12-month period.

During the screening visit, subjects will receive a stool sampling kit and instructions on how and when to collect the stool sample.

Prior to Visit 2, subjects will collect a stool sample and return it to the laboratory with the shipping material provided. At Visit 2 subjects will have blood drawn and urine collected. A stool sampling kit will be dispensed with instructions on how and when to collect the stool sample. Visit 2 must be conducted prior to the start of immunotherapy.

Prior to Visit 3, subjects will collect a stool sample and return it to the laboratory with the shipping material provided. At Visit 3 subjects will have blood drawn and urine collected. A stool sampling kit will be dispensed with instructions on how and when to collect the stool sample.

Prior to Visit 4, subjects will collect a stool sample and return it to the laboratory with the shipping material provided. At Visit 4 subjects will have blood drawn and urine collected. A stool sampling kit will be dispensed with instructions on how and when to collect the stool sample.

Prior to Visit 5, subjects will collect a stool sample and return it to the laboratory with the shipping material provided. At Visit 5 subjects will have blood drawn and urine collected. A stool sampling kit will be dispensed with instructions on how and when to collect the stool sample.

Prior to Visit 6, subjects will collect a stool sample and return it to the laboratory with the shipping material provided. At Visit 6 subjects will have blood drawn and urine collected.

All concomitant medications and adverse events will be recorded. In the event of an adverse event, every effort should be made to collect stool, blood, and urine samples (considered an unscheduled visit).

In the event that a subject discontinues from the study prior to the 12-month visit (Visit 6) all efforts should be made to carry out the assessments for that visit. Visit 6 will also serve as the end of study visit.

Each subject is identified by a unique central identification code that is unique to the study site. This code is only used for study purposes. After informed consent, every person will be given a subject number. The subject code consists of a non interventional study (NIS) code followed by an International Organization for Standardization (ISO) country code, and the subject number. For the duration of the study and afterwards, only the subject's physician will be able to identify the subject based on the subject identification code.

Patient data to be captured in the electronic case report form (eCRF) include demographics, medical history, cancer history, tobacco and alcohol history, diet, prior and concomitant medications, adverse events, and results of tumor scans using the Response Evaluation Criteria in Solid Tumours (iRECIST) criteria.

The trained investigator site staff will enter the data required by the protocol into the eCRFs from source documents (e.g., medical records and study-specific data capture tools as needed) directly into the study database on a central server. All information in the eCRFs must be traceable to these source documents. Data recorded directly into the eCRFs will be defined before study start and the eCRFs will be considered the source data. Clinical Research Associates (CRAs) and a Data Manager will review eCRFs entered by investigational staff for completeness and accuracy. Automatic quality programs check for data discrepancies in the eCRFs and the resulting queries will be notified to the investigational site using an electronic data query process within the Electronic Data Capture (EDC) system. Designated investigator site staff are required to respond to queries and make any necessary changes to the data. Details of the data correction process will be specified in the Data Management Plan. A validated, electronic database will be employed from the EDC system. An audit trail of all changes to this database, including the date, reason for the data change and who made the change, will be maintained within the same database. The audit trail will be part of the archived data at the end of the study.

The complete data management process (data capture, data entry, data validation, checks on plausibility, query handling, data editing after entry, coding, data base closure, etc.) will be defined in advance within a data management plan.

Automatic queries will be defined according to the data management plan. These queries will be auto-generated in the EDC system for data correction and accuracy. Corrections will be entered directly into the system. This procedure will be repeated until all queries are resolved.

The Sponsor will conduct a site visit to verify the qualifications of each investigator, inspect the site facilities, and inform the investigator of responsibilities and the procedures for ensuring adequate and correct documentation. The investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each study participant. All information recorded on the eCRFs for this study must be consistent with the subjects' source documentation (i.e., medical records).

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are ≥ 18 years old who are undergoing any type of cancer immunotherapy
* Subjects who are able to provide written informed consent

Exclusion Criteria:

* Subjects with HIV, Hepatitis B, or Hepatitis C
* Subjects without the mental capacity to complete either a written or online questionnaire, alone or with assistance, or make sound decisions
* Women who are pregnant or who plan on becoming pregnant
* Women who are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person meeting the above criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Checkpoint inhibitor response | 6-12 months
  Response of the tumor to treatment, as evaluated by the iRECIST criteria

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - Bond and Steele Clinic, P.A., Winter Haven, Florida

IPD SHARING:
Plan to Share IPD: No